CLINICAL TRIAL: NCT03513588
Title: A PHASE 1B, RANDOMIZED, DOUBLE-BLIND (SPONSOR-OPEN), PLACEBO-CONTROLLED, PARALLEL GROUP STUDY TO ASSESS THE SAFETY, TOLERABILITY, PHARMACODYNAMICS AND PHARMACOKINETICS OF MULTIPLE ORAL DOSES OF PF- 06865571 FOR 2 WEEKS IN ADULTS WITH NONALCOHOLIC FATTY LIVER DISEASE
Brief Title: 2-Week Study In People With Nonalcoholic Fatty Liver Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: C2541005
Record Dates: First submitted 2018-04-19; First posted 2018-05-01 (Actual); Results first posted 2020-03-13 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2020-02

CONDITIONS: Non-alcoholic Steatohepatitis; Non-alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — ervogastat

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- PF-06865571 100 mg (Experimental)
  Interventions: Drug: PF-06865571
- PF-06865571 600 mg (Experimental)
  Interventions: Drug: PF-06865571

INTERVENTIONS:
Drug: Placebo — tablet, 0 mg, 14 days, every 12 hours
  Arms: Placebo
Drug: PF-06865571 — tablet, 50 mg, 14 days, every 12 hours
  Arms: PF-06865571 100 mg
Drug: PF-06865571 — tablet, 300 mg, 14 days, every 12 hours
  Arms: PF-06865571 600 mg

SUMMARY:
2-week study in people with nonalcoholic fatty liver disease. Study drug at 1 of 2 doses, or placebo, will be given for 14 days. Blood samples, heart monitoring, vital signs, and imaging procedures will be performed.

ELIGIBILITY:
Inclusion Criteria:

* controlled attenuation parameter greater than or equal to 260 dB/m via FibroScan
* liver fat greater than or equal to 6% via MRI

Exclusion Criteria:

* Chronic liver disease
* Type 2 diabetes requiring drug treatment
* Unable to undergo MRI
* History of heart attack or stroke

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-06-21 (Actual); Primary Completion 2019-03-08 (Actual); Study Completion 2019-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (6):
- United States (6):
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - New Haven Clinical Research Unit, New Haven, Connecticut
  - Qps-Mra, Llc, South Miami, Florida
  - PPD Development, LP, Las Vegas, Nevada
  - High Point Clinical Trials Center, High Point, North Carolina
  - Clinical Trials of Texas, Inc., San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Amin NB, Saxena AR, Somayaji V, Dullea R. Inhibition of Diacylglycerol Acyltransferase 2 Versus Diacylglycerol Acyltransferase 1: Potential Therapeutic Implications of Pharmacology. Clin Ther. 2023 Jan;45(1):55-70. doi: 10.1016/j.clinthera.2022.12.008. Epub 2023 Jan 21. PMID 36690550
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C2541005

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received matching placebo tablets orally every 12 hours (Q12H) for 14 days.
- PF-06865571 50 mg: Participants received PF-06865571 50 mg tablets orally Q12H for 14 days.
- PF-06865571 300 mg: Participants received PF-06865571 300 mg tablets orally Q12H for 14 days.
Period: Overall Study
Arm/Group | Placebo | PF-06865571 50 mg | PF-06865571 300 mg
Started | 16 | 17 | 15
Completed | 15 | 15 | 13
Not Completed | 1 | 2 | 2
Not completed — Lost to Follow-up | 0 | 1 | 1
Not completed — Study dosing paused by sponsor | 1 | 1 | 0
Not completed — Death | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least 1 dose of study treatment (PF-06865571 or placebo).
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | PF-06865571 50 mg | PF-06865571 300 mg | Total
Number analyzed (Participants) | 16 | 17 | 15 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.8 (10.5) | 47.0 (8.0) | 48.3 (5.5) | 47.0 (8.2)
Age, Customized [Count of Participants; unit: Participants]
  18-44 years | 7 | 4 | 3 | 14
  45-64 years | 9 | 13 | 12 | 34
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 3 | 13
  Male | 11 | 12 | 12 | 35
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 13 | 14 | 9 | 36
  Black or African American | 3 | 2 | 4 | 9
  Asian | 0 | 1 | 1 | 2
  American Indian or Alaska Native | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Relative Change From Baseline in Whole Liver Fat at Day 15 as Assessed by Magnetic Resonance Imaging (MRI) - Proton Density Fat Fraction (PDFF)
Description: MRI-PDFF is an established method that enables quantification of fat content in the liver. The value of whole liver fat as assessed by MRI-PDFF is expressed in percentage and ranges from 0 to 100% with higher values representing higher liver fat level.
Time Frame: Baseline (Day 1), Day 15
Population: All randomized participants who received at least 1 dose of study treatment (PF-06865571 or placebo) and had whole liver fat assessed at Day 15.
Measure: Least Squares Mean (80% Confidence Interval); unit: percentage of whole liver fat
Arm/Group | Placebo | PF-06865571 50 mg | PF-06865571 300 mg
Number analyzed (Participants) | 15 | 15 | 15
percentage of whole liver fat | -10.94 [-16.65 to -4.83] | -32.62 [-37.02 to -27.90] | -41.14 [-44.91 to -37.12]
Statistical Analysis 1: Comparison: Placebo vs PF-06865571 50 mg; Test type: Other; p < 0.001, ANCOVA; Least Squares Mean Difference = -24.34, 80% CI 2-sided [-31.28 to -16.70]
Statistical Analysis 2: Comparison: Placebo vs PF-06865571 300 mg; Test type: Other; p < 0.001, ANCOVA; Least Squares Mean Difference = -33.91, 80% CI 2-sided [-39.78 to -27.47]

2. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study treatment without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; life-threatening (immediate risk of death); initial or prolonged inpatient hospitalization; persistent or significant disability/incapacity; congenital anomaly/birth defect. Treatment-emergent AEs were those with initial onset or increasing in severity on or after the first dose of investigational product administration. AEs included both SAEs and non-serious AEs.
Time Frame: From first dose of study treatment up to 28-35 days after last dose (maximum of up to 49 days)
Population: All randomized participants who received at least 1 dose of study treatment (PF-06865571 or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-06865571 50 mg | PF-06865571 300 mg
Number analyzed (Participants) | 16 | 17 | 15
Participants
  AEs | 2 | 12 | 9
  SAEs | 0 | 0 | 1

3. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities
Description: Following laboratory parameters were assessed against pre-defined abnormality criteria: hematology (hemoglobin, hematocrit, erythrocytes, mean corpuscular volume, mean corpuscular hemoglobin, mean corpuscular hemoglobin concentration, platelets, leukocytes, lymphocytes, neutrophils, basophils, eosinophils, monocytes); chemistry (total bilirubin, direct bilirubin, indirect bilirubin, aspartate aminotransferase, alanine aminotransferase, gamma glutamyl transferase, alkaline phosphatase, protein, albumin, urea nitrogen, creatinine, urate, sodium, potassium, calcium, chloride, bicarbonate); urinalysis (urine glucose, ketones, urine protein, urine hemoglobin, urobilinogen, urine bilirubin, nitrite, urine erythrocytes, urine leukocytes, hyaline casts); biomarker (total cholesterol, low-density and high-density lipoprotein cholesterol, triglycerides, fasting glucose). Participants with any of the laboratory test abnormalities were counted.
Time Frame: From first dose of study treatment up to 7-10 days after last dose (maximum of up to 24 days)
Population: All randomized participants who received at least 1 dose of study treatment (PF-06865571 or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-06865571 50 mg | PF-06865571 300 mg
Number analyzed (Participants) | 16 | 17 | 15
Participants | 5 | 8 | 6

4. Secondary Outcome: Number of Participants With Vital Sign Abnormalities
Description: Vital sign categorical summarization criteria: 1) supine systolic blood pressure (SBP) <90 millimeters of mercury (mmHg); 2) supine diastolic blood pressure (DBP) <50 mmHg; 3) pulse rate <40 or >120 beats per minute (bpm); 4) change from baseline (increase or decrease) in supine DBP greater than or equal to (>=) 20 mmHg; 5) change from baseline (increase or decrease) in supine SBP >=30 mmHg.
Time Frame: From first dose of study treatment up to 7-10 days after last dose (maximum of up to 24 days)
Population: All randomized participants who received at least 1 dose of study treatment (PF-06865571 or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-06865571 50 mg | PF-06865571 300 mg
Number analyzed (Participants) | 16 | 17 | 15
Participants
  Supine SBP <90 mm Hg | 0 | 0 | 0
  Supine SBP increase >=30 mm Hg | 2 | 1 | 2
  Supine SBP decrease >=30 mm Hg | 1 | 1 | 0
  Supine DBP <50 mmHg | 0 | 0 | 0
  Supine DBP increase >=20 mm Hg | 2 | 0 | 3
  Supine DBP decrease >=20 mm Hg | 1 | 1 | 2
  Pulse rate <40 bpm | 0 | 0 | 0
  Pulse rate >120 bpm | 0 | 0 | 0

5. Secondary Outcome: Number of Participants With Electrocardiogram (ECG) Abnormalities
Description: ECG categorical summarization criteria: 1) QRS interval (time from ECG Q wave to the end of the S wave corresponding to ventricle depolarization): >=140 milliseconds (msec), >=50% change from baseline; 2) PR interval (the interval between the start of the P wave and the start of the QRS complex, corresponding to the time between the onset of the atrial depolarization and onset of ventricular depolarization): >=300 msec, >=25% change when baseline is > 200 msec or >=50% change when baseline is less than or equal to (<=) 200 msec; 3) QTcF interval (heart rate corrected QT [time between the start of the ECG Q wave and the end of the T wave in the heart's electrical cycle] using Fridericia's formula): absolute value of >450 to 480 msec, >480 to 500 msec, >500 msec; a change from baseline of >30 to 60 msec or >60 msec.
Time Frame: From first dose of study treatment up to 7-10 days after last dose (maximum of up to 24 days)
Population: All randomized participants who received at least 1 dose of study treatment (PF-06865571 or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-06865571 50 mg | PF-06865571 300 mg
Number analyzed (Participants) | 16 | 17 | 15
Participants
  PR interval >=300 msec | 0 | 0 | 0
  %Change in PR interval >=25/50% | 0 | 0 | 0
  QRS interval >=140 msec | 0 | 0 | 0
  %Change in QRS interval >=50% | 0 | 0 | 0
  QTcF >450 to <=480 msec | 0 | 0 | 0
  QTcF >480 to <=500 msec | 0 | 0 | 0
  QTcF >500 msec | 0 | 0 | 0
  QTcF change >30 to <=60 msec | 0 | 1 | 1
  QTcF change >60 msec | 0 | 0 | 0

6. Secondary Outcome: Maximum Plasma Concentration (Cmax) For PF-06865571
Description: Cmax of PF-06865571 on Day 14 was observed directly from data. Geometric coefficients of variations were reported as percentages.
Time Frame: Day 14 pre-dose, and 1, 2, 3, 4, 6, 8, 12 hours post-dose
Population: All randomized participants who received at least 1 dose of PF-06865571 (50 mg or 300 mg) and had Cmax data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | PF-06865571 50 mg | PF-06865571 300 mg
Number analyzed (Participants) | 16 | 15
nanograms per milliliter (ng/mL) | 345.5 (35) | 2001 (28)

7. Secondary Outcome: Area Under the Plasma Concentration-Time Profile Over the Dosing Interval (AUCtau) For PF-06865571
Description: AUCtau of PF-06865571 on Day 14 was obtained by linear/log trapezoidal method. The dosing interval (tau) was 12 hours. Geometric coefficients of variations were reported as percentages.
Time Frame: Day 14 pre-dose, and 1, 2, 3, 4, 6, 8, 12 hours post-dose
Population: All randomized participants who received at least 1 dose of PF-06865571 (50 mg or 300 mg) and had AUCtau data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour per milliliter (ng*hr/mL)
Arm/Group | PF-06865571 50 mg | PF-06865571 300 mg
Number analyzed (Participants) | 15 | 15
nanograms*hour per milliliter (ng*hr/mL) | 1036 (35) | 7798 (26)

8. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) For PF-06865571
Description: Tmax of PF-06865571 on Day 14 was observed directly from data as time of Cmax occurrence.
Time Frame: Day 14 pre-dose, and 1, 2, 3, 4, 6, 8, 12 hours post-dose
Population: All randomized participants who received at least 1 dose of PF-06865571 (50 mg or 300 mg) and had Tmax data.
Measure: Median (Full Range); unit: hours
Arm/Group | PF-06865571 50 mg | PF-06865571 300 mg
Number analyzed (Participants) | 16 | 15
hours | 2.00 [1.00 to 4.00] | 2.00 [2.00 to 4.00]

9. Secondary Outcome: Minimum Plasma Concentration (Cmin) For PF-06865571
Description: Cmin of PF-06865571 on Day 14 was observed directly from data. Geometric coefficients of variations were reported as percentages.
Time Frame: Day 14 pre-dose, and 1, 2, 3, 4, 6, 8, 12 hours post-dose
Population: All randomized participants who received at least 1 dose of PF-06865571 (50 mg or 300 mg) and had Cmin data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-06865571 50 mg | PF-06865571 300 mg
Number analyzed (Participants) | 15 | 15
ng/mL | 6.609 (75) | 57.79 (68)

10. Secondary Outcome: Apparent Oral Clearance (CL/F) For PF-06865571
Description: CL/F of PF-06865571 on Day 14 was calculated as Dose/AUCtau. Geometric coefficients of variations were reported as percentages.
Time Frame: Day 14 pre-dose, and 1, 2, 3, 4, 6, 8, 12 hours post-dose
Population: All randomized participants who received at least 1 dose of PF-06865571 (50 mg or 300 mg) and had CL/F data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters per hour (L/hr)
Arm/Group | PF-06865571 50 mg | PF-06865571 300 mg
Number analyzed (Participants) | 15 | 15
liters per hour (L/hr) | 48.30 (35) | 38.49 (26)

11. Secondary Outcome: Peak-to-Trough Ratio (PTR) For PF-06865571
Description: PTR of PF-06865571 on Day 14 was calculated as Cmax/Cmin. Geometric coefficients of variations were reported as percentages.
Time Frame: Day 14 pre-dose, and 1, 2, 3, 4, 6, 8, 12 hours post-dose
Population: All randomized participants who received at least 1 dose of PF-06865571 (50 mg or 300 mg) and had Cmax and non-zero Cmin data for PTR evaluation.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio of concentrations
Arm/Group | PF-06865571 50 mg | PF-06865571 300 mg
Number analyzed (Participants) | 14 | 15
ratio of concentrations | 53.17 (68) | 34.63 (75)

ADVERSE EVENTS:
Time Frame: From first dose of study treatment up to 28-35 days after last dose (maximum of up to 49 days)
Description: The same event may appear as both an AE and an SAE. However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as non-serious in another participant, or 1 participant may have experienced both a serious and non-serious event during the study.
Arm/Group | Placebo | PF-06865571 50 mg | PF-06865571 300 mg
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/17 | 1/15
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/17 | 1/15
Other Adverse Events (participants affected / at risk) | 2/16 | 12/17 | 8/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=16) | PF-06865571 50 mg (N=17) | PF-06865571 300 mg (N=15)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=16) | PF-06865571 50 mg (N=17) | PF-06865571 300 mg (N=15)
Fatigue (General disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 6 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 2
Excessive cerumen production (Ear and labyrinth disorders) | 0 | 0 | 1
Eye pruritus (Eye disorders) | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 2
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Blood pressure increased (Investigations) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 3 | 1
Nervousness (Psychiatric disorders) | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Flushing (Vascular disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2018-02-27): https://cdn.clinicaltrials.gov/large-docs/88/NCT03513588/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-17): https://cdn.clinicaltrials.gov/large-docs/88/NCT03513588/SAP_001.pdf